CLINICAL TRIAL: NCT00429000
Title: Reducing the Prevalence of Hypothermia Among Newborns by Means of Continuous Temperature Monitoring Using Thermospot.
Brief Title: Perinatal Hypothermia, Risk Factors and Long-Term Consequences in Guinea-Bissau, Westafrica
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bandim Health Project (Other)
Collaborators: Lundbeck Foundation (Other); Augustinus Fonden (Other); Danida Travel Grant, (Unknown); Dir E Danielsen og Hustrus Fond, (Unknown); Jakob og Olga Madsens Fond (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007HT
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2007-01-30 (Estimated); Status verified 2007-01

CONDITIONS: Hypothermia; Morbidity; Mortality
Keywords: Hypothermia; Infant mortality; Infant morbidity; Intervention; Randomisation; Longitudinal research.; Low-income country
MeSH Terms: conditions — Hypothermia; Infant Death

INTERVENTIONS:
Device: thermospot

SUMMARY:
Low body temperature (hypothermia (HT)) at birth contributes to infant mortality in low-income countries. A study from Guinéa-Bissau indicates that HT results in an increased mortality rate, which persist at least two months after birth. Therefore interventions that reduce the prevalence of HT might have a significant effect on infant mortality. The purpose of the proposed study is to identify risk factors for HT in an in-hospital setting in Guinea-Bissau and to investigate whether continuous temperature-monitoring enabling early detection of HT and treatment can prevent HT <34,5°C.

DETAILED DESCRIPTION:
Hypothermia (HT) has been recognized as a significant contributor to perinatal morbidity and mortality. Newborns are at risk of developing HT, as their temperature regulation is limited and HT remains a problem in developing countries with poor health care resources, as sub-optimal care for newborns increases the risk of HT. In a longitudinal combined hospital and community study of nearly 3,000 births in Guinea-Bissau we found 8% with HT <34,5°C and that HT within 12 hours of birth is associated with an excess mortality that exists beyond the neonatal period and probably exerts its effects to at least two months of age. The study indicates that the contribution of HT on infant mortality might be higher than presently estimated. In order to meet the fourth goal of The Millennium Developmental Goals, which commits the international community to reducing the mortality in children aged younger then 5 years by two-thirds between 1990 and 2015, a reduction in neonatal mortality rate is essential. Reducing the prevalence of HT might contribute to this. The purpose of the proposed study is to identify risk factors for HT in an in-hospital setting in Guinea-Bissau, and to investigate whether continuous temperature-monitoring enabling early detection of HT and treatment can prevent HT <34,5°C.

The randomised clinical trail will be carried out at the Maternity ward of the National Simão Mendes hospital in Bissau, Guinea Bissau, West Africa. Newborns will be randomised to either standard temperature measurement within the first 12 hours of birth or to continuous temperature monitoring by means of a thermospot, a liquid crystal thermometer shaped as a small small smiley, which changes colour from a green smiling face to black, when the temperature falls below 35.5°C enabling early detection of HT. As it is well known that drying, wrapping and physical contact can improve thermal balance of the newborn, a general intervention aimed at all newborns to prevent HT including changes in existing routines during delivery and immediate perinatal care according to the WHO guidelines will be introduced. All children will benefit from this general intervention. Prior to the intervention study a course in basic neonatology will be held in order to raise awareness of hypothermia among the staff at the maternity. A project assistant will visit all included children in order to follow up on morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Children born at the Maternity ward of the National Simão Mendes hospital in Bissau with a birth weight above 2500g resident within with a predefined geographic area.

Exclusion Criteria:

* Late abortions
* Stillbirths
* Birth weight below 2500g
* Residence within the study area of the Bandim Health Project, as these children are enrolled in other randomised trails.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 788
Dates: Start 2007-01; Study Completion 2007-10

PRIMARY OUTCOMES:
o The prevalence of HT in each group

SECONDARY OUTCOMES:
o Morbidity
o Mortality
o The incidence of infectious diseases
o The prevalence of an adequate response to routine childhood vaccinations
o Frequency of hospital admissions and consultations at local health care centres

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project; Morten Sodemann, PhD, MD, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Bissau Region, Guinea-Bissau